CLINICAL TRIAL: NCT03207763
Title: A Study to Evaluate the Safety, Reactogenicity, and Acceptability of a Placebo Microneedle Patch in Healthy Infants and Young Children
Brief Title: Microneedle Patch Study in Healthy Infants/Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Micron Biomedical, Inc (Industry)
Responsible Party: Principal Investigator, Evan Anderson, Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB00096635
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Vaccination; Skin Absorption
Keywords: Safety; Reactogenicity; Acceptability; Microneedle patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Participating infants and children will receive Microneedle Formulation 1. At least 4 infants or children must complete Day 8 without halting criteria having been met before subjects will be enrolled into the next younger age group within a Cohort. At least the first 2 children will have a microneedle patch initially applied to the skin overlying the shoulder blade. If this site is well tolerated without halting criteria having been met additional microneedle patches may be applied to the same participants and in subsequent participants to the upper arm, forearm, wrist and/or thigh.
  Interventions: Device: Microneedle Formulation 1
- Cohort 2 (Experimental): Participating infants and children will receive Microneedle Formulation 2. At least 4 infants or children must complete Day 8 without halting criteria having been met before subjects will be enrolled into the next younger age group within a Cohort. At least the first 2 children will have a microneedle patch initially applied to the skin overlying the shoulder blade. If this site is well tolerated without halting criteria having been met additional microneedle patches may be applied to the same participants and in subsequent participants to the upper arm, forearm, wrist and/or thigh.
  Interventions: Device: Microneedle Formulation 2

INTERVENTIONS:
Device: Microneedle Formulation 1 — Microneedle patches will be made of solid conical structures made of water-soluble excipients that from the Food and Drug Administration's Generally Recognized as Safe (GRAS) list and/or on the FDA list of inactive ingredients in approved products. The total mass of excipients delivered by placebo microneedle patch will be <1.5 mg. The adhesive backing component is made from hypoallergenic material (commercial medical tapes designed to adhere to skin).
  Microneedle patches will be administered topically by manual application to the skin. The sites of microneedle patch application will be cleaned with an alcohol swab and allowed to dry before the microneedle patch is applied. The microneedle patches will be packaged and provided as single patches.
  Arms: Cohort 1
Device: Microneedle Formulation 2 — Microneedle patches will be made of solid conical structures made of water-soluble excipients that from the Food and Drug Administration's Generally Recognized as Safe (GRAS) list and/or on the FDA list of inactive ingredients in approved products. The ratio of the excipients and excipients used will vary slightly from Formulation 1. The total mass of excipients delivered by placebo microneedle patch will be <1.5 mg. The adhesive backing component is made from hypoallergenic material (commercial medical tapes designed to adhere to skin).
  Microneedle patches will be administered topically by manual application to the skin. The sites of microneedle patch application will be cleaned with an alcohol swab and allowed to dry before the microneedle patch is applied. The microneedle patches will be packaged and provided as single patches.
  Arms: Cohort 2

SUMMARY:
Microneedles can be prepared as a low-cost patch that is simple for patients to apply for vaccine delivery targeting the many antigen-presenting cells present in the skin. Data regarding the safety, reactogenicity, tolerability, and acceptability of a microneedle patch in children are lacking. The goal of this study is to evaluate the safety, reactogenicity, and acceptability of placement of a placebo microneedle patch to the skin of children.

DETAILED DESCRIPTION:
Available vaccine delivery methods include intramuscular or subcutaneous injection are limited by patient needle phobia and the need for trained medical personnel. Alternative routes of vaccination that avoid hypodermic needles have previously been poorly immunogenic, require live vaccines, utilize bulky devices and/or are unsuitable for self-administration. Novel vaccine delivery methods such as microneedles can render vaccination easier and more acceptable to the public by simplifying vaccine access. Microneedles are micron-scale needles that administer vaccine directly into the skin using a simple minimally invasive approach without generating sharps waste. This study is designed to investigate the safety, reactogenicity, and acceptability of a placebo microneedle patch in children.

ELIGIBILITY:
Inclusion Criteria:

* Legally Authorized Representative (LAR) provides written informed consent prior to any study procedures being performed.
* Subject is between the ages of 6 weeks and 24 months, inclusive, on the day of signing informed consent.
* Subject is in good health as determined by vital signs, medical history, and a targeted physical examination.
* LAR is able to understand and comply with required study procedures.

Exclusion Criteria:

* Subject has an acute illness with fever (temperature >100.4 °F) within 72 hours prior to enrollment.
* Subject has a known chronic medical problem.
* Subject has known immunosuppression due to underlying illness or treatment, including (but not limited to): Human Immunodeficiency Virus (or birth to a HIV-positive mother), hepatitis B or C; organ transplant; active cancer or any history of hematologic cancer; receipt of chemotherapy or radiation therapy; congenital immunodeficiency, anatomical or functional asplenia.
* Subject has used long-term* high-dose** oral or parenteral glucocorticoids, or high-dose inhaled steroids.***

  * Long term is defined as taken for 2 weeks or more in total at any time during the past 2 months.

  ** High dose defined as prednisone ≥ 20 mg total daily dose, or equivalent dose of other glucocorticoids.

  *** High dose defined as >800 mcg/day of beclomethasone dipropionate or equivalent.
* Subject has a history of an underlying skin condition (e.g., eczema, atopic dermatitis) or an open lesion (e.g., laceration, abrasion), scar, or rash in the areas of the planned microneedle patch administration which will interfere with the assessment of reactogenicity.
* Subject or family members have a history of keloid formation.
* Subject has any condition that, in the opinion of the investigator, may put the subject at increased risk of harm, may cause the subject to be unable to meet the requirements or might otherwise interfere with evaluations required by the study.
* Subject has received any experimental products within 30 days before study entry or plan to receive experimental products at any time during the study.
* Subject has received a vaccine within 7 days of enrollment or plans to receive a vaccine within 7 days after enrollment.
* Subject has previously received immunoglobulin or blood products.

Ages: 6 Weeks to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Anderson, MD, Principal Investigator — Emory University
Locations (1):
- Emory Children's Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the Emory Children's Center in Atlanta, Georgia. Enrollment began on July 11, 2017 and all follow up was complete by May 15, 2019.
Groups:
- Cohort 1: Participating infants and children receiving Microneedle Formulation 1. Children had a microneedle patch initially applied to the skin overlying the shoulder blade. If the first patch was well tolerated without halting criteria having been met, participants could opt to have two additional microneedle patches applied to the upper arm, forearm, wrist and/or thigh.
- Cohort 2: Participating infants and children receiving Microneedle Formulation 2. Children had a microneedle patch initially applied to the skin overlying the shoulder blade. If the first patch was well tolerated without halting criteria having been met, participants could opt to have two additional microneedle patches applied to the upper arm, forearm, wrist and/or thigh.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 25
Eligible and Opted for Patches 2 and 3 | 5 | 23
Completed Patches 2 and 3 Study | 5 | 23
Completed (Completed follow up for the main study of application of Patch 1) | 7 | 25
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 25 | 33
Age, Customized [Count of Participants; unit: Participants]
  6 weeks to 4 months old | 0 | 10 | 10
  5 to 11 months old | 1 | 8 | 9
  12 to 24 months old | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 5 | 16 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 8 | 20 | 28
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 10 | 15
  White | 1 | 12 | 13
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 25 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Placebo Microneedle Patch-related Serious Adverse Events (SAE).
Description: To evaluate safety following application of the patch topically, microneedle patch-related serious adverse events were recorded. Information collected included event description, date of onset, severity and date of resolution/stabilization of the event. Severity and relationship to study product was assessed by the Investigator or sub-investigator.
Time Frame: Day 1 through the Final Study Visit (Day 27 - 38)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 25
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Grade 3 Placebo Microneedle Patch-related Solicited Adverse Events (AE).
Description: The occurrence of Grade 3 solicited adverse events related to the placebo microneedle patch was recorded. Solicited adverse events were irritability (fussiness), lethargy (drowsiness), decreased appetite, vomiting, and fever. The severity of these adverse events was graded on a scale from 0 to 3 where 0 = not present and 3 = significant, preventing daily activity or a fever of >102.1 degrees Fahrenheit (F).
Time Frame: Up to Day 8 for Patch 1, Day 8 to Day 15 if received Patches 2 and 3
Population: The memory aid to log solicited adverse events was not returned for one participant in Cohort 1 receiving the first patch. The memory aid was not returned for two participants in Cohort 1 receiving the second and third patches.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Patch 1: Participating infants and children receiving Patch 1 of Microneedle Formulation 1
- Cohort 1, Patches 2 and 3: Participating infants and children receiving Patches 2 and 3 of Microneedle Formulation 1
- Cohort 2, Patch 1: Participating infants and children receiving Patch 1 of Microneedle Formulation 2.
- Cohort 2, Patches 2 and 3: Participating infants and children receiving Patches 2 and 3 of Microneedle Formulation 2.
Arm/Group | Cohort 1, Patch 1 | Cohort 1, Patches 2 and 3 | Cohort 2, Patch 1 | Cohort 2, Patches 2 and 3
Number analyzed (Participants) | 7 | 3 | 25 | 23
Participants
  Significant irritability | 0 | 0 | 0 | 1
  Significant lethargy | 0 | 0 | 0 | 0
  Significantly decreased appetite | 0 | 0 | 0 | 0
  Significant vomiting | 0 | 0 | 0 | 0
  Fever >102.1 F | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Application Site Reactogenicity Events.
Description: The occurrence of solicited reactogenicity events at the application site was recorded. The solicited reactogenicity events are reactions that are common or expected to occur with application of a microneedle patch and include induration/swelling, erythema, ecchymosis, itching, pain, and tenderness. The Legally Authorized Representatives (LARs) of participants were provided with a memory aid, thermometer and ruler to record the presence of solicited symptoms and oral temperature. Reactogenicity event details were collected via review of the subject's memory aid and by interview with the subject LAR. Reactogenicity events were graded on a scale from 0 (not present) to 3 (significant or severe).
Time Frame: Up to Day 8 for Patch 1, Day 8 to Day 15 if received Patches 2 and 3
Population: Memory aids were not returned for one participant in Cohort 1 for Patch 1 and two participants in Cohort 1 receiving Patches 2 and 3.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Patch 2: Participating infants and children receiving Patch 2 of Microneedle Formulation 1
- Cohort 1, Patch 3: Participating infants and children receiving Patch 3 of Microneedle Formulation 1
- Cohort 2, Patch 2: Participating infants and children receiving Patch 2 of Microneedle Formulation 2.
- Cohort 2, Patch 3: Participating infants and children receiving Patch 3 of Microneedle Formulation 2.
Arm/Group | Cohort 1, Patch 1 | Cohort 1, Patch 2 | Cohort 1, Patch 3 | Cohort 2, Patch 1 | Cohort 2, Patch 2 | Cohort 2, Patch 3
Number analyzed (Participants) | 7 | 3 | 3 | 25 | 23 | 23
Participants
  Induration/swelling Grade 0 (absent) | 7 | 3 | 3 | 25 | 23 | 23
  Erythema Grade 0 (absent) | 6 | 3 | 3 | 25 | 23 | 23
  Erythema Grade 1 (mild) | 1 | 0 | 0 | 0 | 0 | 0
  Ecchymosis Grade 0 (absent) | 7 | 3 | 3 | 25 | 23 | 23
  Itching Grade 0 (absent) | 6 | 3 | 3 | 25 | 23 | 23
  Itching Grade 1 (mild) | 1 | 0 | 0 | 0 | 0 | 0
  Pain Grade 0 (absent) | 6 | 3 | 3 | 25 | 23 | 23
  Pain Grade 1 (mild) | 1 | 0 | 0 | 0 | 0 | 0
  Tenderness Grade 0 (absent) | 6 | 3 | 3 | 25 | 23 | 23
  Tenderness Grade 1 (mild) | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Grade 3 Placebo Microneedle Patch-related Unsolicited Adverse Events
Description: Grade 3, patch-related unsolicited adverse events (AEs) were recorded. An adverse event is graded as Grade 3 if the event is significant or prevents daily activity.
Time Frame: Day 1 through the Final Study Visit (Day 27 - 38)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 25
Participants | 0 | 0

5. Secondary Outcome: Number of New-onset Medical Conditions (NOMC)
Description: The number of new-onset medical conditions (NOMC) were recorded. NOMC were tabulated by overall and treatment related events.
Time Frame: Day 1 through the Final Study Visit (Day 27 - 38).
Measure: Number; unit: new-onset medical conditions
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 25
new-onset medical conditions | 0 | 0

6. Secondary Outcome: Acceptability of Vaccination Methods
Description: LARs were asked to state their preference for different methods of vaccine delivery, assuming that a vaccine patch were to be available in the next two years. LARs reported their preference for their child receiving 1) a vaccine by shot or nasal spray given by a healthcare worker, 2) a vaccine patch given by a healthcare worker, 3) a vaccine patch given by the LAR but monitored by a healthcare worker, or 4) a vaccine patch given by the LAR at home. LARs rated their preference on a scale from 0 (definitely not) to 10 (definitely so).
Time Frame: Final Visit (Day 27 - 38)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 25
units on a scale
  Shot or spray by healthcare worker | 7.1 (2.5) | 4.8 (4.1)
  Patch by healthcare worker | 8.4 (1.8) | 9.4 (1.2)
  Patch by LAR monitored by healthcare worker | 8.1 (1.7) | 6.8 (3.6)
  Patch by LAR at home | 6.1 (2.9) | 6.0 (3.7)

7. Secondary Outcome: Overall Experience
Description: LARs were asked to report their overall experience with the study so far at each study visit related to Patch 1. Experiences were rated on a scale from 1 to 5 where 1 = very negative and 5 = very positive.
Time Frame: Day 1, Day 2, Day 8, Final Visit (Day 27-38)
Population: The population in this analysis includes LARs who completed this question of the study visit survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 25
units on a scale
  Patch 1, Day 1 | 4.6 (0.5) | 4.5 (0.6)
  Patch 1, Day 2 | 4.6 (0.5) | 4.6 (0.5)
  Patch 1, Day 8 | 4.5 (0.5) | 4.6 (0.7)
  Patches 2 and 3, Day 8: number analyzed (Participants) | 5 | 23
  Patches 2 and 3, Day 8 | 4.2 (1.3) | 4.4 (0.8)
  Patches 2 and 3, Day 9: number analyzed (Participants) | 5 | 22
  Patches 2 and 3, Day 9 | 4.4 (0.9) | 4.7 (0.6)
  Patches 2 and 3, Day 15: number analyzed (Participants) | 5 | 22
  Patches 2 and 3, Day 15 | 4.4 (0.5) | 4.7 (0.5)
  All patchesFinal Visit (Day 27-38): number analyzed (Participants) | 4 | 25
  All patchesFinal Visit (Day 27-38) | 4.5 (0.6) | 4.8 (0.4)

ADVERSE EVENTS:
Time Frame: Data collection for adverse events began at the first study visit and continued through the Final Study Visit, which was a follow up telephone call on Day 27-38.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/25
Other Adverse Events (participants affected / at risk) | 4/8 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=25)
Bug bite (Infections and infestations) | 1 | 0
Teething (Gastrointestinal disorders) | 2 | 0
Bacterial ear infection (Ear and labyrinth disorders) | 1 | 0
Papular rash around site of prior microneedle patch (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperpigmented and macular rash at site of prior microneedle patch (Skin and subcutaneous tissue disorders) | 1 | 0
Viral gastroenteritis (Gastrointestinal disorders) | 0 | 2
Cold symptoms of viral illness (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03207763/Prot_SAP_000.pdf